CLINICAL TRIAL: NCT03970551
Title: Lower Body Muscle Pre-activation in Initial Orthostatic Hypotension: Effects on Orthostatic Tolerance
Brief Title: Lower Body Muscle Pre-activation in Initial Orthostatic Hypotension
Acronym: IOH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Calgary (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: REB19-0792
Record Dates: First submitted 2019-05-24; First posted 2019-05-31 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Orthostatic Intolerance; Syncope; Fainting; Presyncope
Keywords: Initial Orthostatic Hypotension; IOH; Physical Counter-maneuver; Refractory Period; Active Stand; Muscle Tensing; Leg Crossing; Lower Body Muscle Tensing
MeSH Terms: conditions — Orthostatic Intolerance; Syncope | interventions — Exercise Test

STUDY DESIGN:
Intervention Model Description: There will be 6 stands that will involve standing from a sitting position and performing physical counter-maneuvers or a stress test either prior to or following the stand. The order of the interventions will be randomized. Both healthy participants and IOH patients will perform all stands.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- No Physical Intervention (No Intervention): The participant will actively stand up from a seated position without performing any physical counter-maneuvers either prior to or following the stand.
- Supine Knee Raises (Experimental): The participant will perform 30 seconds of raising their knees to their chest while sitting down before actively standing.
  Interventions: Other: Physical Counter-maneuver
- Leg Crossing (Experimental): The participant will actively stand and then immediately cross their legs and tense their leg muscles for 60 seconds.
  Interventions: Other: Physical Counter-maneuver
- Cold Pressor Test (Experimental): The participant will submerge their hands in ice water for approximately 45 seconds.
  Interventions: Other: Stress Test
- Serial 7's Stress Test (Experimental): The participant will perform a mental arithmetic stress test for 30 seconds prior to standing.
  Interventions: Other: Stress Test
- Functional Electrical Stimulation (Experimental): The participant will have their quadriceps passively contracted using mild electrical stimulation for approximately 30 seconds prior to standing.
  Interventions: Other: Functional Electrical Stimulation

INTERVENTIONS:
Other: Physical Counter-maneuver — Physical counter-maneuver targeted at minimizing the large drop in BP seen in IOH patients.
  Arms: Leg Crossing; Supine Knee Raises
Other: Stress Test — Stress test involving submerging your hand in ice water or performing mental arithmetic to increase sympathetic activity.
  Other Names: Cold Pressor Test, Serial 7's Stress Test
  Arms: Cold Pressor Test; Serial 7's Stress Test
Other: Functional Electrical Stimulation — A mild electrical stimulus to passively induce a leg muscle contraction with minimal sympathetic activation.
  Arms: Functional Electrical Stimulation

SUMMARY:
This study is aimed primarily at providing a simple and effective form of treatment to reduce the symptoms of Initial Orthostatic Hypotension (IOH) and prevent syncope. We will first characterize the physiology of IOH, and then we will study four sit-to-stand maneuvers, each with a different stress tests to identify the role of sympathetic activity vs. simple muscle contraction in IOH. Then we will complete an additional two sit-to-stands with interventions designed to decrease the blood pressure drop (and hopefully symptoms) with initial stand. These consist of physical counter maneuvers, which may be a possible treatment that can be used to mitigate the drop in blood pressure (BP) seen in IOH during a stand and relieve presyncope symptoms.

DETAILED DESCRIPTION:
IOH is a form of orthostatic intolerance defined by a transient decrease in systolic blood pressure (SBP) by 40mmHg or diastolic blood pressure (DBP) by 20mmHg within the first 15-30 seconds of assuming a standing position from a supine or seated position. IOH commonly occurs in teenagers and young adults and is associated with presyncope symptoms such as nausea, light-headedness, and blurred vision and may sometimes lead to full syncope. These symptoms are a consequence of cerebral hypoperfusion caused by a rapid reduction in BP and are often present only during an active stand, and not with a passive tilt-table test. This suggests that a muscle activation reflex may play an important role underlying IOH. Identifying the refractory period of leg muscle activation will allow future investigators to accurately determine a common baseline seated period to allow hemodynamic recovery in patients after a stand. This will allow investigators to observe the physiological effects of repeated stands without any interference from a prior stand.

Upon standing there is a large shift of blood (approximately 500 mL) towards the lower extremities and abdomen. With this shift there is a decrease in venous return which results in a drop in BP. Subsequently, the decrease in BP activates the baroreceptors to increase sympathetic activity and reduce parasympathetic activity, which functions to restore BP by increasing heart rate (HR) and total peripheral resistance (TPR).

The underlying physiological mechanism behind the large decrease in blood pressure upon standing in IOH patients has not yet been confirmed. The most widely accepted explanation at this time involves rapid vasodilation localized to the contracting leg muscles during a stand. Research in both human and animal models from the past couple of decades have shown that skeletal muscle resistance vessels can dilate rapidly in response to, as well as in proportion to, a singular brief muscle contraction. This effect may be exaggerated in IOH patients, which could explain the decrease in TPR in IOH patients upon a stand and thus their subsequent drop in blood pressure. Current treatments of IOH include non-pharmacological interventions and physical counter-maneuvers such as standing up slowly or sitting up first before fully standing.

Physical counter-measures function to oppose the gravitational pull experienced on systemic circulation during a stand. During a stand, a large percentage of circulating blood shifts towards the lower extremities and abdomen resulting in blood pooling. Gravitational venous pooling can be minimized and opposed by performing a physical countermeasure such as a lower-body muscle contraction to translocate blood centrally. Sustained tensing of the lower-body muscles prevents further peripheral pooling in the legs and abdomen.

The investigators hypothesize that pre-activation of lower body muscles prior to standing, will attenuate the drop in SBP seen in IOH patients upon a stand, and alleviate symptoms of IOH, compared to an active stand without muscle pre-activation. The study participant will complete 14 active stands in total within a single day. The first 8 stands will be in an attempt to define the refractoriness of leg muscle activation. The next 4 stands will involve stress tests prior to standing to isolate the roles of sympathetic activity vs. simple muscle contraction. The final 2 stands will involve physical counter-maneuvers intended to mitigate the large drop in BP seen in IOH patients upon a stand.

The first 8 stands will be performed from a seated position. They will begin at a 20 minute seated baseline before the first stand, then in a random order perform stands after baseline durations of 30 sec, 2 min, 3 min, 4 min, 5 min, 7 min, and 10 min.

The next 4 stands will also be performed from a seated position. The interventions that will be performed in a random order are: (1) free stand with no intervention, (2) Serial 7's mental arithmetic stress test, (3) Cold Pressor stress test, (4) functional electrical stimulation.

The final 2 stands will be performed from a seated position as well. The interventions that will be performed in a random order are: (1) supine knee raises and tensing prior to standing and (2) leg crossing and tensing after standing. The entire study will take approximately 3-4 hours.

The study participant will be instrumented in a fasting state and on an empty bladder. The investigators will apply skin electrodes to continuously monitor heart rate and record an ECG. BP will be monitored continuously using finger volume clamp photoplethysmography and calibrated with intermittent brachial cuff measurements. From the continuous BP waveform, the investigators can obtain an estimate of stroke volume, cardiac output, and systemic vascular resistance (Modelflow). Oxygen saturation will be assessed from a finger probe. Middle cerebral blood flow velocity will be assessed using transcranial doppler (TCD).

ELIGIBILITY:
Inclusion Criteria:

* Either have initial orthostatic hypotension or are a healthy volunteer
* 18-50 years old
* Male or Female
* Ability to travel to Libin Cardiovascular Institute of Alberta Autonomic Research Testing Lab in the Teaching, Research & Wellness Building at the University of Calgary, Calgary, AB
* Able and willing to provide informed consent

Exclusion Criteria:

* Inability to stand up or perform leg exercises without assistance
* Sustained orthostatic hypotension past 3 minutes of standing
* Pregnant

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Magnitude of change in SBP from sitting to stand with a physical intervention | < 5 minutes
  The magnitude of change in SBP from sitting to stand when the participant performs muscle pre-activation before a stand compared to no intervention at all.

SECONDARY OUTCOMES:
Differences in Vanderbilt Orthostatic Symptoms Score (VOSS) Symptom Rating | < 5 minutes
  Subjective symptom scoring as reported by participant during each study arm. The VOSS evaluates 9 symptoms on a 0 to 10 scale with 0 being no symptom to 10 being worst ever symptom. The total score ranges from 0-90, with a higher score being more severe symptoms.
  The 9 symptoms are mental clouding, blurred vision, shortness of breath, rapid heartbeat, tremulousness, chest discomfort, headache, lightheadedness, and nausea. The participant's VOSS score will be compared across the 4 arms of this study.
  The VOSS score has been previously used in multiple publications
Nadir SBP | < 5 minutes
  Nadir systolic blood pressure when standing during each study arm.
Peak HR | < 5 minutes
  Peak heart rate when standing during each study arm.
Cerebral Blood Flow Velocity (CBFV) | < 5 minutes
  CBFV when standing during each study arm.

CONTACTS AND LOCATIONS:
Overall Officials: Satish R Raj, MD, MSCI, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No
I will not be sharing individual participant data.

REFERENCES:
- [Background] da Silva RM. Syncope: epidemiology, etiology, and prognosis. Front Physiol. 2014 Dec 8;5:471. doi: 10.3389/fphys.2014.00471. eCollection 2014. PMID 25538626
- [Background] McJunkin B, Rose B, Amin O, Shah N, Sharma S, Modi S, Kemper S, Yousaf M. Detecting initial orthostatic hypotension: a novel approach. J Am Soc Hypertens. 2015 May;9(5):365-9. doi: 10.1016/j.jash.2015.02.006. Epub 2015 Feb 13. PMID 25816712
- [Background] Eser I, Khorshid L, Gunes UY, Demir Y. The effect of different body positions on blood pressure. J Clin Nurs. 2007 Jan;16(1):137-40. doi: 10.1111/j.1365-2702.2005.01494.x. PMID 17181675
- [Background] Wieling W, Krediet CT, van Dijk N, Linzer M, Tschakovsky ME. Initial orthostatic hypotension: review of a forgotten condition. Clin Sci (Lond). 2007 Feb;112(3):157-65. doi: 10.1042/CS20060091. PMID 17199559
- [Background] Stewart JM, Clarke D. "He's dizzy when he stands up": an introduction to initial orthostatic hypotension. J Pediatr. 2011 Mar;158(3):499-504. doi: 10.1016/j.jpeds.2010.09.004. No abstract available. PMID 20970148
- [Background] Stewart JM. Mechanisms of sympathetic regulation in orthostatic intolerance. J Appl Physiol (1985). 2012 Nov;113(10):1659-68. doi: 10.1152/japplphysiol.00266.2012. Epub 2012 Jun 7. PMID 22678960
- [Background] Tschakovsky ME, Matusiak K, Vipond C, McVicar L. Lower limb-localized vascular phenomena explain initial orthostatic hypotension upon standing from squat. Am J Physiol Heart Circ Physiol. 2011 Nov;301(5):H2102-12. doi: 10.1152/ajpheart.00571.2011. Epub 2011 Aug 19. PMID 21856921
- [Background] Wieling W, van Dijk N, Thijs RD, de Lange FJ, Krediet CT, Halliwill JR. Physical countermeasures to increase orthostatic tolerance. J Intern Med. 2015 Jan;277(1):69-82. doi: 10.1111/joim.12249. Epub 2014 May 5. No abstract available. PMID 24697914
- [Background] Krediet CT, Go-Schon IK, Kim YS, Linzer M, Van Lieshout JJ, Wieling W. Management of initial orthostatic hypotension: lower body muscle tensing attenuates the transient arterial blood pressure decrease upon standing from squatting. Clin Sci (Lond). 2007 Nov;113(10):401-7. doi: 10.1042/CS20070064. PMID 17561808
- [Background] van Twist DJL, Dinh T, Bouwmans EME, Kroon AA. Initial orthostatic hypotension among patients with unexplained syncope: An overlooked diagnosis? Int J Cardiol. 2018 Nov 15;271:269-273. doi: 10.1016/j.ijcard.2018.05.043. PMID 30223355
- [Derived] Sheikh NA, Phillips AA, Ranada S, Lloyd M, Kogut K, Bourne KM, Jorge JG, Lei LY, Sheldon RS, Exner DV, Runte M, Raj SR. Mitigating Initial Orthostatic Hypotension: Mechanistic Roles of Muscle Contraction Versus Sympathetic Activation. Hypertension. 2022 Mar;79(3):638-647. doi: 10.1161/HYPERTENSIONAHA.121.18580. Epub 2022 Jan 6. PMID 34990207